CLINICAL TRIAL: NCT05202405
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover, Phase 1 Study to Evaluate the Safety and Pharmacokinetics of AD-221 Compared to Coadministration of AD-221A and AD-221B in Healty Adult Volunteers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of AD-221 Compared to Coadministration of AD-221A and AD-221B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-221PK
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-01

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1 : Reference Drug(AD-221A and AD-221B) Period 2 : Test Drug(AD-221)
  Interventions: Drug: AD-221; Drug: AD-221A and AD-221B
- Sequence B (Experimental): Period 1 : Test Drug(AD-221) Period 2 : Reference Drug(AD-221A and AD-221B)
  Interventions: Drug: AD-221; Drug: AD-221A and AD-221B

INTERVENTIONS:
Drug: AD-221 — AD-221 Oral Tablet
Drug: AD-221A and AD-221B — AD-221A Oral Tablet + AD-221B Oral Tablet

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-221 in healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety profiles of AD-221 compared with coadministration AD-221A and AD-221B in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | pre-dose to 72 hours
  Cmax of AD-221
Area Under the Curve in time plot (AUCt) | pre-dose to 72 hours
  AUCt of AD-221

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song J, Bae S, Yu KS, Lee S. Comparison of pharmacokinetics of a fixed-dose combination of atorvastatin/ezetimibe 5 mg/10 mg versus separate tablets in healthy subjects. Transl Clin Pharmacol. 2025 Mar;33(1):40-49. doi: 10.12793/tcp.2025.33.e5. Epub 2025 Mar 24. PMID 40206873